CLINICAL TRIAL: NCT02909569
Title: Relieving Chronic Itch : Oral Medication
Brief Title: Relieving Chronic Itch: Oral Medication
Acronym: CIPS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Contract could not be agreed on.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP9110
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Pruritis
MeSH Terms: conditions — Pruritus | interventions — INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB039110 (Experimental): INCN039110 400 mg QD for 20 weeks. Subjects without clinical response after four weeks will increase to 600mg QD.
  Interventions: Drug: INCB039110

INTERVENTIONS:
Drug: INCB039110 — All subjects will receive 400 mg PO QD for 12 weeks. If no clinical response after four weeks, dose will be increased to 600 mg PO QD. Total duration of subject participation will be six study visit over 20 weeks.

SUMMARY:
This study evaluates the effect of twice daily dose of INCB39110 in the treatment of itch in adults.

DETAILED DESCRIPTION:
Chronic idiopathic itch accompanies low-grade skin inflammation. These inflammatory features are associated with cytokine production which signal through the common JAK1-STAT pathway. It is therefore theorized that a selective JAK1 inhibitor such as INCB039110 may provide relief of itch symptom.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female subjects aged 18 years or older
* Diagnosed with chronic idiopathic pruritus (CIP) with an NRS Itch Score of ≥ 7 at both Screening and Baseline
* Diagnosis of CIP for at least 6 weeks prior to screening
* Willingness to avoid pregnancy or fathering of children
* Ability and willingness to provide written informed consent
* Willing and able to comply with all study requirements and restrictions
* Willing to not participate in any other interventional trial for the duration of their participation
* Subjects must be in good health as determined by medical history, physical examination, electrocardiogram, clinical laboratory tests and vital signs
* Failure of a course 2-week course of treatment with topical triamcinolone 0.1% ointment BID
* Histopathological demonstration of skin dermal edema, eosinophils, mast cell activation or lymphocytic infiltration

Exclusion Criteria:

1. Chronic pruritus due to a defined primary dermatologic disorder (e.g., atopic dermatitis, psoriasis, etc.)
2. Patients with a prior diagnosis of excoriation disorder
3. Use of topical treatments for CIP (other than bland emollients) within 1 week of baseline
4. Systemic immunosuppressive or immunomodulating drugs (eg, oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolat mofetil, azathioprine) within 4 weeks of baseline
5. Subjects with cytopenias at screening, defined as:

   1. Leukocytes < 3 × 109/L
   2. Neutrophils < lower limit of normal
   3. Lymphocytes < 0.8 × 109/L
   4. Hemoglobin < 10 g/dL
   5. Platelets < 100 × 109/L
6. Unwilling or unable to follow medication restrictions or unwilling or unable to sufficiently washout from use of restricted medication
7. Use of any prohibited medications (see Section 5.8) within 14 days or 5 half-lives (whichever is longer) of the baseline visit
8. Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal gastrointestinal, endocrine or metabolic dysfunction unless currently controlled and stable, including (but not limited to) the following:

   1. Positive for hepatitis C antibody test (anti-HCAbF) with detectable RNA
   2. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb);
   3. Positive for HIV (DUO test, p24 antigen)
9. Active malignancy
10. Subjects with a history of malignancy, except for the following adequately treated, nonmetastatic malignancies: basal cell skin cancer, squamous cell carcinomas of the skin, or in situ cervical cancer
11. History (including family history) or current evidence of congenital long QT syndrome or known acquired QT prolongation
12. Exposure to any investigational medication, including placebo, within 60 days of the Baseline Visit
13. History of intolerance and/or hypersensitivity to medications similar to INCB039110 (e.g., Xeljanz)
14. Participation in a previous INCB39110 trial
15. Subjects with severely impaired liver function (Child-Pugh Class C) or end-stage renal disease on dialysis or at least 1 of the following:

    1. Serum creatinine > 1.5 mg/dL;
    2. Alanine aminotransferase or aspartate aminotransferase ≥ 1.5 × upper limit of normal
16. Anyone affiliated with the site or sponsor and/or anyone who may consent under duress
17. Any other sound medical reason as determined by the Investigator including any condition which may lead to an unfavorable risk-benefit of study participation, may interfere with study compliance or may confound study results
18. Subjects taking potent systemic CYP3A4 inhibitors or fluconazole within 2 weeks or 5 half-lives, whichever is longer, before the baseline visit
19. Subjects who have previously received JAK inhibitors, systemic or topical (e.g. ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib and pacritinib)
20. Women who were pregnant or breastfeeding within 4 months before screening.
21. Current or recent history (< 30 days before screening and/or < 45 days before randomization) of a clinically meaningful bacterial, fungal, parasitic, or mycobacterial infection
22. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy or uncontrolled hypertension (blood pressure > 150/90 mmHg) unless approved by medical monitor/sponsor
23. History of alcoholism or drug addiction within 1 year before screening, or current alcohol or drug use that, in the opinion of the investigator, will interfere with the subject's ability to comply with the administration schedule and study assessments
24. Subjects who have received systemic chemotherapy at any time
25. Subjects who anticipate receiving a live or live-attenuated vaccination from screening through the final follow-up visit
26. Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the administration schedule and study evaluations

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) itch score | Baseline to 12 weeks
  Absolute change from Baseline NRS itch score to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kim, MD/MTR, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No